CLINICAL TRIAL: NCT04646811
Title: TRI-FR : Multicentric Randomized Evaluation of Tricuspid Valve Percutaneous Repair System (Clip for the Tricuspid Valve) in the Treatment of Severe Secondary Tricuspid Disorders
Brief Title: Evaluation of Tricuspid Valve Percutaneous Repair System in the Treatment of Severe Secondary Tricuspid Disorders
Acronym: TRI-FR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC18_8851_TRI-FR; 2020-A00645-34 (Other: N° IDRCB)
Record Dates: First submitted 2020-11-10; First posted 2020-11-30 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Tricuspid Regurgitation
Keywords: secondary Tricuspid Regurgitation; least severe Tricuspid Regurgitation; symptomatic patients
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tricuspid valve (Experimental): tricuspid valve percutaneous repair strategy with clip for the tricuspid valve
  Interventions: Procedure: Tricuspid valve
- Best medical treatment (Other)
  Interventions: Other: Best medical treatment

INTERVENTIONS:
Procedure: Tricuspid valve — Clip for the tricuspid valve implantation on top of best medical therapy
  Arms: Tricuspid valve
Other: Best medical treatment — Best medical therapy alone
  Arms: Best medical treatment

SUMMARY:
Tricuspid regurgitation (TR) is a long-overdue valvular pathology. Its prevalence is significant and increasing with the aging of the population. It is often a consequence of chronic left cardiac pathologies or atrial fibrillation. Surgical treatment is recommended in severe symptomatic TR or when the tricuspid annulus is dilated with TR identified prior to scheduled left heart valve surgery. TR are mainly secondary (complicating left heart disease, pulmonary hypertension, atrial fibrillation and atrial dilatation) and pose a difficult problem related to the prognosis. The risk of death or hospitalization is high under medical treatment. Nevertheless, the surgical results are disappointing with significant morbidity and mortality, which are increased by associated comorbidities that are frequent in these sorts of patients. The benefit-risk assessment of surgery is limited by multiple confounders.

This justifies the evaluation of alternative methods aimed at correcting TR with less interventional risk.

The Clip for the tricuspid valve has been evaluated in the TRILUMINATE trial (inclusion of 85 patients with moderate-to-severe symptomatic TR with a 6-month follow-up). The Triclip system appears to be safe and effective at reducing tricuspid regurgitation by at least one grade. This reduction could translate to significant clinical improvement at 6 months post-procedure. It justified the European Conformity (CE) mark obtention.

A very similar system for the mitral valve (Mitraclip) was previously tested in the randomized EVEREST II study against conventional surgery. The results of the EVEREST II trial justified the recourse to percutaneous edge-to edge mitral repair in patients with primary mitral regurgitation when the patient is contraindicated to conventional surgery.

The Mitra-FR study made it possible to study the role of Mitraclip for treating patient suffering from a secondary mitral insufficiency. It leads to the implementation of this technique in selected patients.

For secondary TR, several series underscored its prevalence and its clinical consequences. TR treatment justifies the proposal for a randomized study. As a matter of fact, evidence for treating are seriously lacking. Surgical surveys report hospital mortality ~ 8.8%. It, therefore, seems necessary to conduct a study as robust as possible to evaluate the contribution of clip for the tricuspid valve (as an innovative percutaneous technique) compared to conventional pharmacological treatment in patients who are unsuitable for a surgical isolated correction of the TR and who has suitable anatomy for clip for the tricuspid valve. It will be necessary to demonstrate clinical, functional (quality of life), echocardiographic and biological benefit of the percutaneous treatment vs optimized medical treatment alone.

DETAILED DESCRIPTION:
The principal objective is to demonstrate, over a period of 12-month after randomization, that, on the Packer composite clinical endpoint (CCS) (combining NYHA class, patient global assessment (PGA) and major cardio-vascular events), the tricuspid valve percutaneous repair strategy with clip for the tricuspid valve is superior to best (optimized) medical treatment (BMT) in symptomatic patients with at least severe secondary TR. The Packer clinical composite score is eventually a three-level ordered categorical endpoint, each randomized patient being classifying as improved, unchanged, or worsen, depending on the clinical response over the follow-up period and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

Pre-Inclusion Criteria:

1. Age ≥ 18 years
2. Symptomatic secondary (at least) severe TR (Carpentier Type IIIB (restrictive) and / or I (tricuspid annulus dilation)) stable for at least 30 days
3. NYHA functional class II to IV without cirrhosis and/or ascites
4. Signs of heart failure in the previous 12-months with or without having been hospitalized
5. Stable optimized medical and/or interventional treatment
6. Ineligible for corrective action on the valve by surgical approach after a specialized multidisciplinary consultation ("heart team") including at least a cardio-thoracic surgeon, an interventional cardiologist, an imaging-cardiologist and an Anesthesiologist).
7. Signature of an informed consent

   Definitive Inclusion Criteria:
8. Central core-laboratory analysis : TR characterized before Implantation by at least one of the following criteria:

   * Regurgitation volume > 45 mL / beat
   * Surface of the regurgitant orifice > 40 mm²
   * Vena contracta> 7mm
   * Gap between leaflets ≤ 10 mm (at the presumed location of the clip)

Then after the TR severity grading; the Clinical eligibility Committee will valid the inclusion.

Non Inclusion Criteria:

1. Patient treated with Mitraclip or other percutaneous approach on the mitral valve in the past 3-month
2. Any prior tricuspid valve procedure that would interfere with placement of the Triclip device
3. Tricuspid valve leaflet anatomy which may preclude clip implantation, proper clip positioning on the leaflets or sufficient reduction in TR. This may include:

   * Tricuspid valve anatomy not evaluable by TTE and TEE
   * Active endocarditis
   * Evidence of calcification in the grasping area
   * Evidence of stenosis (mean pressure gradient > 5 mmHg or surface area ≤1cm²
   * Presence of a severe coaptation defect (> 1cm) of the tricuspid leaflets
   * Severe leaflet defect(s) preventing proper device placement
   * Epstein anomaly - identified by having a normal annulus position while the valve leaflets are attached to the walls and septum of the right ventricle
4. Myocardial infarction or coronary bypass surgery in the past 3-month
5. Left ventricular ejection fraction ≤35%
6. Cardiac Resynchronization therapy for less than 3-month and patients having a TR that is clearly related to the right ventricular lead positioning
7. Cardioversion for less than 6 weeks
8. Life expectancy irrespective of the valvular heart disease <1 year (due to co-morbidities)
9. Other scheduled cardiac surgery (including registration in cardiac transplant list)
10. Coronary angioplasty in the preceding month
11. Current infection requiring prescription of antibiotics
12. End-stage renal failure (dialysis patient)
13. Severe hepatic insufficiency (disruption of liver metabolism associated with coagulation disorders (factor V <50%))
14. Stroke in the previous 3-month
15. Uncontrolled pre- capillary pulmonary hypertension (right catheterization required) (systolic pulmonary pressure > 60 mmHg)
16. Tricuspid prosthetic valve
17. Pace maker lead or ICD lead that would prevent appropriate placement of the Triclips
18. Nitinol allergy
19. Contraindication, allergy or hypersensibility to dual anti-platelet and anticoagulant therapy
20. Ongoing infection requiring antibiotic therapy
21. Evidence of intra vascular or intra cardiac thrombus
22. Patient who are included in another research protocol
23. Protected person (adults legally protected (under judicial protection, guardianship or supervision), person deprived of their liberty, pregnant woman, lactating woman and minor)
24. Absence of coverage by a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Milton Packer clinical composite score | 12 months
  Milton Packer clinical composite score classifies each patient into 1 of 3 categories (improved, worsened, unchanged), and is determined aggregating evaluation functional using NYHA class, quality of life score using patient global assessment and number of major cardio-vascular events

SECONDARY OUTCOMES:
number of participants with all-cause mortality | 12 months
number of participants with tricuspid valve surgery | 12 months
rate of heart failure hospitalizations | 12 months
assessment of quality of life improvement | 0 and 12 months
  Kansas City Cardiomyopathy Questionnaire score (KCCQ) The responses are categorized under 3 subscales (symptom burden, physical limitation and quality of life) with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The total KCCQ score represents the mean of the three subscale scores.
quality of life score | 6 and 12 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) The responses are categorized under 3 subscales (symptom burden, physical limitation and quality of life) with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The total KCCQ score represents the mean of the three subscale scores.
quality of life score | 6 and 12 months
  Minnesota Living with Heart Failure (MLHF)
quality of life score | 6 and 12 months
  EQ5D-5L The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system :
  5 dimensions : mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
  5 levels : no problems,slight problems, moderate, problems and extreme. Each level corresponds to 1 digit number. The digits for the 5 dimensions are combined into a 5-digit number.
  The EQ VAS : on a vertical visual analogue scale, 100 'The best health you can imagine' 0 'The worst health you can imagine'.
quality of life score | 6 and 12 months
  Patient global assessment (PGA)
functional evaluation | 6 and 12 months
  NYHA functional class
severity of the Tricuspid Regurgitation (TR) | 6 and 12 months
  TR grade
walking distance | 6 and 12 months
  6-minute walk test
echocardiography parameters | 6 and 12 months
  right heart function
echocardiography parameters | 6 and 12 months
  right heart cavities sizes
echocardiography parameters | 6 and 12 months
  degree of tricuspid regurgitation
echocardiography parameters | 6 and 12 months
  stenosis
biological parameters | 6 and 12 months
  parameters renal : creatinine, clearance, AST
biological parameters | 6 and 12 months
  hepatic function
biological parameters | 6 and 12 months
  NT-proBNP
overall survival | 6 and 12 months
number of cardiovascular death | 6 and 12 months
number of major cardiovascular events | 6 and 12 months
Incremental Cost-Effectiveness Ratio expressed as cost per QALY | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Donal Erwan, Principal Investigator — CHU Rennes
Locations (26):
- Belgium (3):
  - Service de Cardiologie AZ Sint-Jan, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - CHU Liège, Liège
- France (23):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Bordeaux - Hôpital Cardiologique du Haut-Lévêque, Bordeaux
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHU Lille, Lille
  - Hôpital Privé Le Bois, Lille
  - Hospices Civils de Lyon Groupement Hospitalier EST, Lyon
  - APHM - Hôpital La Timone, Marseille
  - Hôpital de Saint-Joseph, Marseille
  - Institut Cardiovasculaire Paris Sud Hôpital Jacques Cartier, Massy
  - Clinique du Millénaire, Montpellier
  - CHU Nantes - Hôtel Dieu et Hôpital Nord Laennec, Nantes
  - Hôpital Bichat, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - Centre Cardiologique du Nord, Saint-Denis
  - CHU La Réunion, Saint-Denis
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Toulouse - Hôpital Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - CHU Tours - Hôpital Trousseau, Tours
  - Médipôle Lyon-Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coisne A, L'Official G, Dreyfus J, Ternacle J, Leurent G, Le Roux PY, Ganivet A, Sportouch-Dukhan C, Lavie-Badie Y, Guerin P, Rouleau F, Diakov C, Van Der Heyden J, Obadia JF, Nejjari M, Karam N, Bernard A, Neylon A, Pierrard R, Tchetche D, Ghostine S, Istratoaie S, Donal E. Echocardiographic Outcomes After Transcatheter Edge-to-Edge Repair in Patients With Isolated Tricuspid Regurgitation: The Tri.Fr Trial. JACC Cardiovasc Imaging. 2025 Nov 18:S1936-878X(25)00531-5. doi: 10.1016/j.jcmg.2025.09.010. Online ahead of print. PMID 41258847
- [Derived] Donal E, Dreyfus J, Leurent G, Coisne A, Leroux PY, Ganivet A, Sportouch C, Lavie-Badie Y, Guerin P, Rouleau F, Diakov C, van der Heyden J, Lafitte S, Obadia JF, Nejjari M, Karam N, Bernard A, Neylon A, Pierrard R, Tchetche D, Ghostine S, Ducrocq G, Si Moussi T, Jeu A, Peltier M, Cosyns B, Le Dolley Y, Habib G, Auffret V, Le Ven F, Picard F, Piriou N, Laperche T, Galli E, Istratoaie S, Jouan J, Bonnet G, de Groote P, Anselmi A, Trochu JN, Oger E; Tri-Fr Investigators. Transcatheter Edge-to-Edge Repair for Severe Isolated Tricuspid Regurgitation: The Tri.Fr Randomized Clinical Trial. JAMA. 2025 Jan 14;333(2):124-132. doi: 10.1001/jama.2024.21189. PMID 39602173
- [Derived] Donal E, Leurent G, Iung B. Are We Right to Believe in the Value of Transcatheter Treatment of Secondary Tricuspid Regurgitation? J Am Coll Cardiol. 2021 Jan 26;77(3):240-242. doi: 10.1016/j.jacc.2020.11.037. No abstract available. PMID 33478647